CLINICAL TRIAL: NCT05389358
Title: Pilot Intervention for Addressing Intimate Partner Violence, Mental Health, and HIV in Antenatal Care
Brief Title: Addressing Intimate Partner Violence, Mental Health, and HIV in Antenatal Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Abigail Hatcher, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K01MH12118501; M210216; 5K01MH121185 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Partner Abuse; Depression; Adherence, Medication
Keywords: intimate partner violence; perinatal depression; ART adherence; HIV; antenatal care; prevention of mother-to-child transmission
MeSH Terms: conditions — Depression; Medication Adherence | interventions — Referral and Consultation; Poliovirus Vaccine, Inactivated; Mental Health

STUDY DESIGN:
Intervention Model Description: 2 primary health clinics offering antenatal care services in inner-city Johannesburg, South Africa will be randomized to receive intervention or enhanced standard of care. Within each clinic n=40 participants will take part in baseline, midline, and endline assessments.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants at routine antenatal care will not know whether their clinic is the intervention or enhanced usual care arm, since both will offer support that is over-and-above standard care. Outcomes will be assessed using self-completed tablet computers, so there is no outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Asiphephe (meaning "Let us stay safe") intervention is a problem-solving therapy manual delivered in a one-on-one setting by lay health workers during routine antenatal care. Lay health workers are already employed by the Department of Health and are trained in-service (30 hours) and receive monthly supervision (total of approximately 6 one-on-one hours; 15 group hours). Asiphephe includes illustrated job aids, participant workbook, intervention checklist, and an intervention manual. The model is informed by problem-solving therapy (Lund, 2018), trauma-informed coping (Sikkema, 2018) and safety planning (Garcia-Moreno, forthcoming) and was piloted with 12 health workers with input from 3 global mental health experts.
  Interventions: Behavioral: Asiphephe health worker training; Behavioral: Asiphephe therapeutic sessions; Other: IPV assessment; Other: Referral for IPV or Mental Health
- Enhanced standard of care (Active Comparator): The enhanced standard of care condition will entail a clinic-wide training (5 hours) on IPV, mental health, and HIV care in order to sensitize staff to the nature of the research. The clinic will receive access to established referral network to which participants can gain additional help with violence exposure or mental ill health. Participants in this arm will also be observed for adverse events and social harms, with referrals made appropriately by study staff.
  Interventions: Other: IPV assessment; Other: Referral for IPV or Mental Health

INTERVENTIONS:
Behavioral: Asiphephe health worker training — Lay health workers are already employed by the Department of Health and are trained in-service (30 hours) and receive monthly supervision (total of approximately 6 one-on-one hours; 15 group hours).
  Arms: Intervention
Behavioral: Asiphephe therapeutic sessions — Asiphephe sessions are manualized using illustrated job aids, a participant workbook, session checklists, and an intervention manual. The model is informed by problem-solving therapy (Lund, 2018), trauma-informed coping (Sikkema, 2018) and safety planning (Garcia-Moreno, forthcoming) and was piloted with 12 health workers with input from 3 global mental health experts.
  Arms: Intervention
Other: IPV assessment — IPV intensity as measured by WHO Multicountry Study Instrument at a cut-off of any past-year physical/sexual/psychological violence exposure vs. none
Other: Referral for IPV or Mental Health — Study staff are trained to recognize signs or symptoms of distress and to make appropriate referrals to appropriate community-based services, if necessary. Experienced mental health professionals on the investigative can be consulted or referred to should a participant exhibit severe symptom of mental distress.

SUMMARY:
This quasi-experimental feasibility study recruit n=40 participants from each of two public antenatal clinics in Johannesburg, South Africa. Using the Bowen et al. approach, key feasibility study questions will be those around acceptability, implementation, and promising effects on intermediate variable. While this pilot trial is not powered to determine efficacy, it can help establish whether intervention targets the appropriate intermediate mechanisms (i.e. primary endpoints of IPV exposure and depressive symptoms) and moves intended outcomes in the right direction (i.e. towards better adherence as measured by self-reported adherence).

DETAILED DESCRIPTION:
Prevention of mother-to-child transmission (PMTCT) programs are effective if women take medication regularly, yet many perinatal women in sub-Saharan Africa have sup-optimal adherence. Intimate partner violence (IPV) worsens women's ability to adhere to antiretroviral therapy (ART), and leads to higher rates of depression. In a quasi-experimental feasibility study in South Africa, 2 inner-city Johannesburg clinics will be assigned to intervention or enhanced standard of care conditions. Intervention consists of training health workers to deliver one-on-one sessions in pregnancy (4 sessions) and postpartum (2 sessions) using problem-solving therapy and safety planning. Following n=80 women in a prospective cohort will allow for preliminarily assessment of intervention effects on: perinatal depression, IPV exposure, and ART adherence at 6 months postpartum. Additional qualitative research with 10 providers and 15 beneficiaries will help us qualitatively assess acceptability of intervention content, measures, and study conditions. This pilot trial can establish acceptability of intervention and control conditions and provide preliminary point estimates to inform future trial design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older (the age of research consent in South Africa)
* currently pregnant and less than 30 weeks gestation (from antenatal green card)
* speak a study language (English, isiZulu, Sesotho)
* living with HIV (self-reported and confirmed on green card)
* report past-year IPV (score of ≥1 on WHO multicountry study instrument)
* are willing to provide informed consent

Exclusion Criteria:

* fail to meet all of the inclusion criteria
* at risk of immediate danger (current suicidality, homicidality, or risk to child safety)
* planning to terminate the pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression | 6 months postpartum
  Depressive symptoms using Patient Health Questionnaire-9 will be assessed as a continuous marker of symptomology (with ≥13 indicating probable depression)
Intimate partner violence | 6 months postpartum
  IPV exposure will be measured using the World Health Organization multicountry study instrument of behaviorally-specific likert-type items about frequency of physical, sexual, or psychological violence from a partner. Any IPV will be defined as an affirmative response to any physical, sexual, or psychological violence question. For primary outcome assessment, the WHO instrument will be examined as a continuous measure summing all standardized response items as a marker of IPV intensity (Tsai, 2016).

SECONDARY OUTCOMES:
ART adherence | 6 months postpartum
  Self-reported ART adherence will be collected using a multi-item measure (Wilson et al, 2014).

OTHER OUTCOMES:
Viral suppression | 6 months postpartum
  Log10 viral load (VL) will be abstracted from medical records.
Anxiety | 6 months postpartum
  Anxiety symptoms will measured by Generalized Anxiety Disorder scale-7 with a cut-off of 8 suggesting probable generalized anxiety.
PTSD | 6 months postpartum
  Post traumatic stress symptoms will be measured by the Harvard Trauma Questionnaire with symptom severity assessed as continuous scale.

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Malvern Clinic, Johannesburg, Gauteng
  - Yeoville Clinic, Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: No
The pilot nature of this study and small sample mean we will not make IDP available to researchers outside of our investigative team.